CLINICAL TRIAL: NCT05237388
Title: Janus Kinase-STAT Inhibition to Reduce APOL1 Associated Kidney Disease
Acronym: JUSTICE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00108755; R01MD016401-01 (NIH)
Record Dates: First submitted 2022-01-31; First posted 2022-02-14 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
Keywords: APOL1; focal segmental glomerulosclerosis (FSGS)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Glomerulosclerosis, Focal Segmental | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baricitinib (Experimental): Participants will take one pill of Baricitinib daily with their regular medications.
  Interventions: Drug: Baricitinib
- Placebo (Placebo Comparator): Participants will take a Baricitinib placebo pill matching Baricitinib daily with their regular medications.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — One pill daily
  Arms: Baricitinib
Drug: Placebo — Baricitinib placebo pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the drug, baricitinib, is safe and effective in reducing high levels of albumin in the urine (albuminuria) in African American/Blacks with APOL1- associated focal segmental glomerulosclerosis (FSGS) and non-diabetic APOL1-associated chronic kidney disease due to hypertension (HTN-CKD).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-70 years
* High Risk APOL1 genotype (i.e., G1G1, G2G2, or G1G2)
* FSGS diagnosed by kidney biopsy or clinically diagnosed HTN-CKD
* UACR ≥300 mg/dL
* Estimated glomerular filtration rate (eGFR) ≥26 ml/min/1.73 m2 at screening
* Stable antihypertensive regimen for ≥ 1 month prior to enrolment
* Able to provide written informed consent

Exclusion Criteria:

* Diabetes
* HIV
* Sickle cell disease.
* Tip variant of FSGS.
* Systolic BP >180 mmHg or diastolic BP >90 mmHg based on average of 3 measurements.
* Active serious viral, bacterial, fungal or parasitic infection.
* Symptomatic herpes zoster infection within 12 weeks prior to study entry.
* Positive hepatitis B surface antigen during screening (could enroll after treatment).
* Previous kidney transplant.
* History of chronic liver disease with the most recent available aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the ULN or the most recent available total bilirubin ≥1.5 times the ULN
* Hemoglobin <10 g/dL.
* Absolute lymphocyte count (ALC)<500cells/mm3 or absolute neutrophil count (ANC) < 1000 cells/mm3.
* Pregnant or nursing at time of enrollment
* Prior or current treatment with JAK inhibitor.
* Current use of potent immunosuppressants such as abatacept, adalimumab, anakinra, azathioprine, certolizumab, etanercept, golimumab, infliximab, probenecid, rituximab, ruxolitinib, sarilumab, tofacitinib, or tocilizumab.
* High dose corticosteroids (>10 mg per day of prednisone or equivalent) or an unstable dosing regimen of corticosteroids within 2 weeks of study entry or within 6 weeks of planned randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in albuminuria (UACR) | Baseline, monthly for 6 months

SECONDARY OUTCOMES:
Percent change in eGFR as measured by blood test | Baseline, monthly for 6 months
Percent change in urine CXCL 9-11 as measured by urine test | Baseline, monthly for 6 months
Number of adverse events as measured by patient report | Up to 6 months
Number of adverse events as measured by clinical lab value of hemoglobin less than 9.5g/dL | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Opeyemi Olabisi, MD, Principal Investigator — Duke University
Locations (1):
- Duke Research at Pickett Road, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No